CLINICAL TRIAL: NCT01128907
Title: Galactomannan Antigen and Real Time - PCR for Aspergillus DNA Detection in Bronchoalveolar Lavage. Application in the Diagnosis of Invasive Aspergillosis in Neutropenic Patients
Brief Title: Galactomannan Antigen in Bronchoalveolar Lavage in the Diagnosis of Invasive Aspergillosis in Neutropenic Patients
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: PR03/03/2007
Record Dates: First submitted 2010-03-19; First posted 2010-05-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Invasive Aspergillosis
Keywords: Invasive Aspergillosis in neutropenic patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Hematological neutropenic patients at high risk of Invasive Aspergillosis with persistent fever and an opportunist infection suspicion.
- 2: Patients without hematological illness and without Invasive Aspergillosis suspicion.

SUMMARY:
Invasive Aspergillosis (IA) is a very serious fungal infection. Hematological patients are the most affected group. IA has a very high morbimortality due to its rapid progression and because it is very difficult to be early diagnosed. Diagnosis is used to be done too late or even post-mortem. They are two new methods (techniques) trying to make the diagnosis on an early stage: detection of Galactomannan antigen of Aspergillus species and real - time polymerase chain reaction (PCR) of its DNA in blood. IA in immunocompromised patients is mainly located in lungs, so our hypothesis is that in patients where the investigators suspect IA the investigators should find earlier Galactomannan antigen or real -time PCR of Aspergillus in respiratory samples such as bronchoalveolar lavage (BAL), and its detection could be useful for diagnosis.

Objectives: To detect Galactomannan Antigen and Real Time - PCR for Aspergillus DNA in bronchoalveolar lavage. To validate the routine utility of these tests in BAL as a diagnostic method of IA and investigate if Galactomannan Antigen and Real Time - PCR for Aspergillus DNA in bronchoalveolar lavage can optimize blood test sensibility.

Methods: Prospective study. The investigators will include 200 patients. 100 of them will be hematological patients, neutropenic and at high risk to develop an IA. The other 100 will be patients without risk or no suspicion at all of IA. The investigators will perform a BAL in all patients. And blood detection of Galactomannan Antigen in hematological patients. The investigators will perform a standard microbiological culture of BAL and Galactomannan Antigen in both samples (bronchoalveolar lavage and blood). The investigators also will carry out Real Time - PCR for Aspergillus DNA detection in bronchoalveolar lavage.

Expected results: To detect Galactomannan Antigen and Real Time - PCR for Aspergillus DNA in BAL with more specificity and making earlier diagnosis than in blood. The investigators also expect to implant these techniques in BAL in the routine for IA diagnosis in neutropenic patients.

ELIGIBILITY:
Inclusion Criteria:

* 100 BAL in hematological neutropenic patients at high risk of IA, admitted to our hospital, in which we usually perform a BAL for microbiological study when they present persistent fever and an opportunist infection suspicion.
* 100 BAL in patients without hematological illness and without IA suspicion, in which we perform an BAL because of another reason.

Exclusion Criteria:

* Patients without fulfilling inclusion criteria.
* Patients with some contraindication to perform a bronchoscopy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. hematological neutropenic patients at high risk of IA in which we usually perform a BAL for microbiological study when they present persistent fever and an opportunist infection suspicion.
  2. patients without hematological illness and without IA suspicion, in which we perform an BAL because of another reason.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2006-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Galactomannan antigen and Real Time - PCR for Aspergillus DNA detection in bronchoalveolar lavage. | 3 years
  Cross-sectional design.

SECONDARY OUTCOMES:
Utility of Galactomannan antigen and Real Time - PCR for Aspergillus DNA in BAL as a diagnostic method of IA. | 3 years
  Cross-sectional design.
Galactomannan Antigen and Real Time- PCR for Aspergillus DNA in bronchoalveolar lavage can optimize blood test sensibility? | 3 years
  cross-sectional design.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain